CLINICAL TRIAL: NCT02016768
Title: Decompressive Cervical Surgery for Antihypertensive Effect in Patients With Cervical Spondylosis and Hypertension-A Cohort Study
Brief Title: Decompressive Cervical Surgery and Hypertension
Status: Completed | Type: Observational
Sponsor: Peking University First Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Hong Liu, Dr., Peking University First Hospital
Other Study IDs: PUCRP201304
Record Dates: First submitted 2013-12-15; First posted 2013-12-20 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Myelopathy, Compressive; Hypertension
MeSH Terms: conditions — Spinal Cord Compression; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- operation: To make decompressive cervical surgery, either anterior cervical discectomy and fusion or posterior laminoplasty on the patients suffering from cervical spondylotic myelopathy and hypertension.
  Interventions: Procedure: decompressive cervical surgery

INTERVENTIONS:
Procedure: decompressive cervical surgery — To make decompressive cervical surgery, either anterior cervical discectomy and fusion or posterior laminoplasty on the patients suffering from cervical spondylotic myelopathy and hypertension.
  Other Names: anterior cervical discectomy fusion; posterior laminoplasty

SUMMARY:
There is a relationship between CSM and hypertension, probably a cause/effect relationship, and investigators term this type of hypertension "cervicogenic hypertension". Abnormally functioning serotonergic pacemaker cells in the dorsal raphe nucleus inappropriately activate and inhibit parts of the central and autonomic nervous systems as part of a chronic stress response, which causes hypertension and migraine. This theory is now being expanded to encompass both CSM and essential hypertension, the idea being that these two conditions are intimately related.

DETAILED DESCRIPTION:
Cervical spondylotic myelopathy (CSM) and hypertension are both very common diseases in the general population.Investigators have also observed previously hypertensive patients with CSM become normotensive following decompressive cervical surgery and no longer need antihypertensive medications. Both observations are difficult to explain according to current theories of the two diseases.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of cervical spondylosis myelopathy
* Be at least 18 years of age
* Office-measured systolic BP≧140mmHg
* Ability to adhere to study protocol
* Have signed an approved informed consent form for participation in this study

Exclusion Criteria:

* Have hypertension secondary to a treatable cause
* Have prior cervical spine surgery
* Are pregnant or contemplating pregnancy during the 3-month follow-up period
* People deny to join the study
* Are unable to comply with protocol requirements
* Are unlikely to survive the protocol follow-up period
* Are enrolled in another concurrent clinical trial
* Visual Analogue Scale≥4

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at our Spine Center suffering signs and symptoms of cervical myelopathy and with evidence of radiographic cervical cord compression with hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in the systolic blood pressure(SBP) measured by 24-hour Ambulatory Blood Pressure Monitoring(ABPM) on 1st month and 3th month post-operation. | twice ABPM prior to operation and 1st month, 3th month post-operation.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, Master, Principal Investigator — Peking Unversity First Hospital
Locations (1):
- Hong LIu, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Liu H, Wang HB, Wu L, Wang SJ, Yang ZC, Ma RY, Reilly KH, Yan XY, Ji P, Wu YF. Effects of decompressive cervical surgery on blood pressure in cervical spondylosis patients with hypertension: a time series cohort study. BMC Surg. 2016 Jan 6;16:2. doi: 10.1186/s12893-015-0117-y. PMID 26738624